CLINICAL TRIAL: NCT07221942
Title: Pembrolizumab Maintenance After Enfortumab Vedotin/Pembrolizumab Induction in Front-Line Metastatic Urothelial Carcinoma
Brief Title: Pembrolizumab Maintenance After Enfortumab Vedotin (EV)/Pembro Induction in Front-Line Metastatic Urothelial Carcinoma
Acronym: IMPROEV
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-1029; GU-229 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2025-10-17; First posted 2025-10-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Urothelial Carcinoma; Unresectable Urothelial Carcinoma; Advanced Urothelial Carcinoma
Keywords: Urothelial carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction EV + Pembrolizumab Followed by Maintenance Pembrolizumab (Experimental): Participants will receive induction therapy with enfortumab vedotin (EV) plus pembrolizumab (P) for 6 cycles (approximately 18 weeks). EV will be administered at 1.25 mg/kg IV on Days 1 and 8 of each 21-day cycle (starting dose of 1 mg/kg allowed), and pembrolizumab at 200 mg IV on Day 1 of each cycle. Patients achieving complete or partial response will transition to maintenance pembrolizumab at 400 mg IV every 6 weeks or 200 mg IV every 3 weeks for up to 2 years. Dose modifications for EV are permitted per protocol; no dose adjustments for pembrolizumab. Treatment continues until disease progression, unacceptable toxicity, or completion of maintenance therapy.
  Interventions: Drug: Enfortumab vedotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Enfortumab vedotin — EV will be administered at 1.25 mg/kg IV on Days 1 and 8 of each 21-day cycle
Drug: Pembrolizumab — Pembrolizumab will be administered at 200 mg IV on Day 1 of each 21-day cycle

SUMMARY:
This is a single-arm, open-label, non-randomized Phase II trial evaluating the efficacy of induction therapy with enfortumab vedotin (EV) plus pembrolizumab (P) for 18 weeks (6 cycles), followed by maintenance pembrolizumab in treatment-naïve patients with metastatic urothelial carcinoma (mUC). Approximately 97 patients will be enrolled. Induction consists of EV (1.25 mg/kg IV on Days 1 and 8 of each 21-day cycle; starting dose of 1 mg/kg allowed) and P (200 mg IV on Day 1 of each cycle). Radiographic assessments occur after 3 and 6 cycles. Patients achieving complete or partial response transition to maintenance P (400 mg IV every 6 weeks or 200 mg IV every 3 weeks) for up to 2 years. Dose modifications for EV are permitted per protocol; no dose adjustments for P. Treatment continues until disease progression, unacceptable toxicity, or completion of maintenance therapy. Patients will enter long-term or survival follow-up as applicable.

DETAILED DESCRIPTION:
This is a single-arm, open-label, non-randomized Phase II trial designed to evaluate the efficacy of induction therapy with enfortumab vedotin (EV) plus pembrolizumab (P) for 18 weeks (6 cycles), followed by maintenance pembrolizumab in treatment-naïve patients with metastatic urothelial carcinoma (mUC). Approximately 97 patients will be enrolled, with recruitment anticipated to begin in 2025.

Induction Phase (18 weeks):

Patients will receive EV (1.25 mg/kg IV on Days 1 and 8 of each 21-day cycle; starting dose of 1 mg/kg allowed per physician discretion) and P (200 mg IV on Day 1 of each cycle). The first radiographic assessment will occur after 3 cycles (approximately 9 weeks). Patients demonstrating clinical benefit (CR or PR per RECIST v1.1) will receive 3 additional cycles of EV/P, followed by a second radiographic assessment after 6 cycles (approximately 18 weeks). Patients achieving CR or PR will transition to the maintenance phase. Patients with stable disease may continue EV/P or transition to maintenance P based on patient/physician discretion. Patients experiencing progression during induction may seek alternative treatments.

Maintenance Phase:

Responding patients (CR/PR) will receive P at 400 mg IV every 6 weeks for up to 2 years, or 200 mg IV every 3 weeks per physician preference. The 2-year duration aligns with the maximum pembrolizumab exposure in EV-302. Radiographic assessments will occur every 12 weeks during maintenance. Patients will continue treatment until disease progression, unacceptable toxicity, or completion of maintenance therapy. Patients progressing on P maintenance may resume EV.

Follow-Up:

Patients will enter Survival Follow-up upon progression or toxicity requiring cessation of therapy. If a patient discontinues one drug due to toxicity or near complete response, they may continue on the other drug and remain on study. Both drugs may be discontinued early for toxicity or near complete response at physician discretion; these patients enter Long-term Follow-up. Patients who resume therapy after early discontinuation remain in Long-term Follow-up until progression, then transition to Survival Follow-up. Patients with suboptimal disease control or progression after EV schedule de-escalation may return to the original EV schedule at the highest tolerated dose per physician discretion. Dose adjustments for EV (1.25 mg/kg → 1 mg/kg → 0.75 mg/kg) are permitted per EV-302 guidelines. No dose adjustments for P will be made. Treatment may be held for up to 8 weeks for toxicity management; if held beyond 8 weeks, patients enter Long-term Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and radiographically confirmed locally advanced, unresectable urothelial carcinoma.
* Patients should not have received prior systemic therapy for metastatic disease.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v1.1
* Patients may have received prior neoadjuvant or adjuvant immune checkpoint inhibitor therapy for localized disease and are eligible if they completed the treatment ≥12 months prior to initiating treatment on this clinical trial.
* ECOG performance status 0-2
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document
* Archival tumor biospecimen (when available) must be procured for correlative evaluation. If tumor tissue is not available or accessible despite good faith efforts, patient may still be treated on study. Formalin fixed, paraffin embedded (FFPE) tissue block(s) or at least 25 unbaked, unstained slides are required. Tissue samples taken from a metastatic lesion prior to the start of screening are acceptable.
* Normal organ and marrow function as defined below.

  * Absolute neutrophil count > 1,000/mm3 unless patient has constitutional neutropenia
  * Platelets > 100,000/µl
  * Hemoglobin > 8.0 g/dL
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x upper limit of normal (ULN) or <3.5 x ULN if liver metastases
  * Creatinine Clearance >20 ml/min

Exclusion Criteria:

* Patients who have received prior monomethyl auristatin E (MMAE)-based antibody-drug conjugates (ADCs) for urothelial cancer.
* Grade 2 or higher baseline sensory or motor neuropathy.
* Uncontrolled diabetes (HbA1c >8%)
* Patients with uncontrolled and untreated central nervous system (CNS) metastases.

  * Prior radiation to CNS metastases is permitted.
  * Prior history of CNS disease that has responded to previous systemic therapy is permitted only if no recurrence.
  * Patient should not have leptomeningeal disease
  * CNS metastases have been clinically stable for at least 6 weeks prior to screening and baseline scans show no evidence of new or enlarged metastasis.
  * If requiring steroid treatment for CNS metastases, the patient is on stable dose < 10 mg/day of prednisone or equivalent for at least 2 weeks prior to starting treatment
* Uncontrolled intercurrent illness including, but not limited to ongoing or active untreated infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would substantially impair the patient's ability to comply with study requirements. Efforts should be made to provide reasonable accommodations before determining exclusion based on social limitations.
* Subjects with a history of another invasive malignancy within 3 years before the first dose of study drug that cannot be watched and requires treatment, or any evidence of residual disease from a previously diagnosed malignancy that cannot be watched and requires treatment. Adjuvant hormonal therapy for breast cancer is allowed.
* Currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of first dose of enfortumab vedotin. Routine antimicrobial prophylaxis is permitted.
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with enfortumab vedotin.
* History of idiopathic pulmonary fibrosis; organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Prior allogeneic stem cell or solid organ transplant.
* Other underlying medical condition that, in the opinion of the investigator, would impair the ability of the patient to receive or tolerate the planned treatment and follow-up; any known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study.
* Patients with active tuberculosis.
* Pregnant or breast feeding
* History of autoimmune diseases. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

  * Patients with vitiligo or residual autoimmune hypothyroidism on stable doses of hormone replacement are permitted to enroll.
  * Patients with type 1 diabetes mellitus (T1DM) on a stable dose of insulin are permitted to enroll.
  * Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* On high dose steroids at the time of study enrollment, defined as >10 mg prednisone (or bioequivalent), including steroids used for management of intracranial lesions. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
* Patients who received prior immunotherapy for mUC or for an alternative malignancy are eligible unless they developed an immune related adverse event while on therapy requiring cessation of therapy or use of disease modifying agents, corticosteroids, or immunosuppressive drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-03 (Estimated)

PRIMARY OUTCOMES:
18-month progression-free survival (PFS) | 18 months
  radiographic progression or death from any cause within 18 months of initiating treatment

SECONDARY OUTCOMES:
Overall Survival (OS) | 4 years
  Time from initiating treatment to death from any cause, to capture long-term survival benefits
Duration of Response (DoR) | 4 years
  Time from first objective response (CR/PR) to radiographic progression or death, providing insight into the sustained efficacy of the treatment
PFS 2 after EV rechallenge | 4 years
  Since patients progressing after completing induction EV/P will be able to receive EV re-challenge, we will measure PFS with EV rechallenge measured from the start of EV rechallenge to the next progression defined by RECIST 1.1 or death
Treatment-free interval | 4 years
  Time from the completion of induction EV/P to either EV re-initiation or the start of another therapy, measuring how long patients remain off treatment
Incidence of Peripheral neuropathy | 4 years
  Changes in neuropathy-related symptoms will be assessed using the EORTC QLQ-CIPN20 survey, which evaluates sensory, motor, and autonomic neuropathy symptoms
Quality of Life (QoL) using EORTC QLQ-C30 (European Organization For Research And Treatment Of Cancer Quality of Life Questionnaire) | 4 years
  Assessed using EORTC QLQ-C30 questionnaire; higher scores indicate better global health status
Quality of Life (QoL) using QLQ-BLM30 | 4 years
  QLQ-BLM30 a disease-specific module designed to assess health-related quality of life in patients with muscle-invasive bladder cancer. Higher scores indicate more symptoms, which means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Ghatalia, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No